CLINICAL TRIAL: NCT04800367
Title: Romosozumab for Premenopausal Idiopathic Osteoporosis
Brief Title: Romosozumab/Denosumab Study for Premenopausal IOP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Adi Cohen, Professor of Medicine at CUIMC, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT1202
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Premenopausal Idiopathic Osteoporosis
Keywords: denosumab; romosozumab; premenopausal osteoporosis
MeSH Terms: interventions — romosozumab; Denosumab

STUDY DESIGN:
Intervention Model Description: 12 months of romosozumab followed by 12 months of denosumab
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Romosozumab followed by denosumab (Experimental): Romosozumab 210 mg subcutaneous injection, once a month for 12 months followed by denosumab 60 mg subcutaneous injection, once every six months for 12 months.
  Interventions: Drug: Romosozumab Prefilled Syringe [Evenity]; Drug: Denosumab 60 MG/ML Prefilled Syringe [Prolia]

INTERVENTIONS:
Drug: Romosozumab Prefilled Syringe [Evenity] — 2 syringes of 105 MG/1.17 mL subcutaneous solution injected one after the other, once a month from study baseline through 11 month visit
  Other Names: Evenity
Drug: Denosumab 60 MG/ML Prefilled Syringe [Prolia] — 1 subcutaneous injection of 60 mg/mL every six months from study 12 month visit through the 24 month visit. Injections occur at the 12 and 18 month visits.
  Other Names: Prolia

SUMMARY:
The overarching goal of the research program is to define optimal treatment for premenopausal women with clinically significant fracture syndromes that require medical therapy. The investigators hypothesize that romosozumab will be associated with improvements in bone mass and microarchitecture in premenopausal women, and also that the responses and response rates will exceed those observed in premenopausal women treated with teriparatide. The investigators will test this hypothesis in this phase 2 study of 30 premenopausal women with idiopathic osteoporosis (IOP) who will receive 12M of romosozumab 210 mg monthly followed by 12M of denosumab 60 mg SC q6M. Aim 1 will define the within-group effects of this regimen. Aim 2 will compare results from participants treated with romosozumab-denosumab to the investigator's well-characterized historical controls treated with teriparatide followed by denosumab.

DETAILED DESCRIPTION:
Romosozumab is an anti-sclerostin antibody that provides powerful skeletal benefits through concomitant osteoanabolic and antiresorptive effects on bone. In postmenopausal women, romosozumab is associated with larger increases in spine and hip BMD in comparison to teriparatide. Romosozumab has an extremely low reported nonresponse rate and transition to denosumab after romosozumab leads to further BMD increases and sustained anti-fracture efficacy.

Therefore, the investigators hypothesize that romosozumab will be associated with improvements in bone mass in premenopausal women, and also that the responses and response rates will exceed those observed in premenopausal women treated with teriparatide. The investigators will test this hypothesis in this phase 2 study of 30 premenopausal women with IOP who will receive 12M of romosozumab 210 mg monthly followed by 12M of denosumab 60 mg SC q6M ("romosozumab-denosumab").

Aim 1 will define the within-group effect of romosozumab-denosumab. The primary outcome variable will be the within-group change in areal BMD by DXA at the lumbar spine at 12M. Secondary outcome variables include change in aBMD by DXA at the total hip, femoral neck and 1/3 radius at 12M and change in aBMD at all sites at 24 months.

Aim 2 will compare results from participants treated with romosozumab-denosumab to the well-characterized historical controls treated with 24 months of teriparatide alone, and a subset of those treated with 24 months of teriparatide followed by 12 months of denosumab. The investigators hypothesize that romosozumab over 12M and romosozumab-denosumab over 24M will be associated with larger BMD gains compared to 12M and 24M of teriparatide. The investigators also hypothesize that 24M of romosozumab-denosumab will be associated with comparable BMD gains vs. historical controls treated with 36M of teriparatide-denosumab.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, aged 18-48, with regular menses and no historical or biochemical secondary cause of osteoporosis; the lower age limit is to ensure epiphyses are fused, the upper to make it less likely that women will enter menopause during the study. All subjects under age 25 will be screened (bone age radiograph) prior to enrollment to rule out open epiphyses.

  * Documented adult fractures judged to be low-trauma (equivalent to a fall from a standing height or less) and T-score or Z-score ≤ -1.5 at the LS, TH or FN.
  * Must agree to use highly effective contraception throughout the period of study drug administration.

Highly effective contraception includes methods considered by the CDC to be >99% effective (e.g. vasectomized partner, tubal ligation, hysterectomy, IUD) as well as a combination of barrier method (condoms) with hormonal contraception considered to be > 90% effective (oral contraceptive pill, patch or ring). Systemic progestin only methods (oral or implanted) are not included due to their effect on systemic estrogen levels and thus potential effects on bone health in this premenopausal population.

Exclusion Criteria:

* Any cardiovascular disease: history of myocardial infarction (MI) or stroke. Normal electrocardiogram (ECG) or ECG with no clinically significant abnormality is required at study entry.
* Conditions requiring chronic anticoagulation (coumadin, heparins)
* Early follicular phase serum FSH>20 mIU/ml (to exclude perimenopausal women)
* Disorders of mineral metabolism: primary/secondary hyperparathyroidism, osteomalacia (including that associated with a diagnosis of hypophosphatasia), vitamin D deficiency

  * Suspicion of osteomalacia (elevated alkaline phosphatase, bone pain exacerbated by weight bearing, bone tenderness)
  * Vitamin D deficiency (serum 25-OHD<30ng/ml). Women with levels of 10-29 ng/ml will be eligible after treatment with vitamin D has resulted in levels ≥30 ng/ml.
  * Hypocalcemia
  * Hypercalciuria: urinary calcium excretion over 300 mg/g Cr that can not be effectively lowered with medical management (reduced calcium intake, thiazide diuretics). As in our prior studies, prevalent nephrolithiasis in the absence of pretreatment hypercalciuria is not an exclusion.
* Current pregnancy or lactation

  * Highly effective contraception is required, pregnancy testing is performed at each visit
* Current active eating disorder, hypothalamic or exercise induced amenorrhea. Patients with past history of these disorders, resolved > 1 year ago, are eligible to participate. The Eating Aptitude Test -Questionnaire is given to identify women with subclinical eating disorders
* Current malignancy
* Endocrinopathy: new onset untreated hyperthyroidism/hypothyroidism, Cushing's syndrome, prolactinoma
* Renal insufficiency (eGFR below 60 ml/min)
* Liver disease (AST, ALT, bilirubin, total alkaline phosphatase activity above upper normal limit)
* Intestinal malabsorption disorders including but not limited to pancreatic insufficiency, active Crohn Disease or untreated celiac disease.
* History/current GCs, anticonvulsants, anticoagulants, methotrexate, GnRH agonists to suppress menstruation
* Oral glucocorticoid dose equivalent >5 mg prednisone for >3 months.
* Current use of specific anticonvulsants (carbamazepine, phenytoin, phenobarbital), methotrexate, GnRH agonists to suppress menstruation. Subjects who completed treatment with these medications > 1 year ago are eligible to participate
* Current GCs (oral GC equivalent to 5mg prednisone or more). Subjects who completed treatment with these medications for ≤ 3 months, > 1 year ago are eligible to participate.
* Current anticoagulant use; past use of warfarin (Coumadin) or low molecular weight heparin is not an exclusion, although known thrombotic disease is an exclusion
* Depo Provera (depot medroxyprogesterone acetate) unless taken after age 20, more than 5 years ago
* Drugs for osteoporosis (raloxifene, bisphosphonates, denosumab, calcitonin, TPTD/abaloparatide): Subjects who discontinue these medications will be eligible:

  * 3 months after stopping raloxifene or calcitonin
  * 12 months after stopping abaloparatide, teriparatide, alendronate, risedronate, ibandronate, or pamidronate
  * 24 months after the last dose of zoledronate
  * 18 months after the last dose of denosumab. Subjects who have received ≤ 6 months of teriparatide or abaloparatide will be eligible 2 months after the last dose.

Subjects who have received ≤ 12 months of teriparatide or abaloparatide will be eligible 6 months after the last dose.

* Women with a history of dental extraction or other invasive dental work within 3 months, or who require invasive dental work within the next two years, will be excluded
* Hypersensitivity to romosozumab or denosumab

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percent change in lumbar spine BMD by DXA | Baseline-12 months
  Within-group percent change in lumbar spine BMD by DXA at 12M

SECONDARY OUTCOMES:
Percent change in lumbar spine BMD by DXA | Baseline, 6 month, 12 month, 18 month, 24 month
  Within-group percent change in lumbar spine BMD every 6 months
Percent change in total hip BMD by DXA | Baseline, 6 month, 12 month, 18 month, 24 month
  Within-group percent change in total hip BMD every 6 months
Percent change in femoral neck BMD by DXA | Baseline, 6 month, 12 month, 18 month, 24 month
  Within-group percent change in femoral neck BMD every 6 months
Percent change in distal radius BMD by DXA | Baseline, 6 month, 12 month, 18 month, 24 month
  Within-group percent change in distal radius BMD every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adi Cohen, MD, Principal Investigator — Columbia University; Elizabeth Shane, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States